CLINICAL TRIAL: NCT04268069
Title: A Phase 2, Multi-center, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy and Safety of PL9643 Ophthalmic Solution Compared to Placebo in Subjects With Dry Eye
Brief Title: Efficacy and Safety of PL9643 Ophthalmic Solution in Subjects With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Collaborators: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL9643-201
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Ophthalmic Solution (vehicle) (Placebo Comparator): vehicle
  Interventions: Drug: Placebo Ophthalmic Solution
- PL9643 Ophthalmic Solution (Active Comparator): PL9643 Ophthalmic Solution
  Interventions: Drug: PL9643 Ophthalmic Solution

INTERVENTIONS:
Drug: PL9643 Ophthalmic Solution — PL9643 Ophthalmic Solution as topical ophthalmic drops administered bilaterally for 12 weeks.
  Arms: PL9643 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Placebo solution as topical ophthalmic drops administered bilaterally for 12 weeks.
  Arms: Placebo Ophthalmic Solution (vehicle)

SUMMARY:
Evaluation of safety and efficacy of PL9643 Ophthalmic Solution compared to placebo for the treatment of the signs and symptoms of dry eye.

DETAILED DESCRIPTION:
The clinical trial is a Phase 2, multi center, randomized, double masked and placebo controlled study.

During a 14-day study run-in period (for the purpose of subject selection) prior to randomization, all subjects will receive Placebo Ophthalmic Solution (vehicle) bilaterally. During the screening period, exposure to the CAE® will be conducted to ascertain eligibility to enter the study at Visit 1 and Visit 2. Those who qualify at Visit 2 will be randomized to receive study drug in a double-masked fashion for 12 weeks. The CAE® exposure will occur at all Visits.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Provided written informed consent.
* Have a reported history of dry eye
* Have a history of use or desire to use eye drops for dry eye symptoms
* Have corrected visual acuity greater than or equal to +0.7 in both eyes

Exclusion Criteria:

* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal)
* Have any planned ocular and/or lid surgeries over the study period.
* Have an uncontrolled systemic disease.
* Be a woman who is pregnant, nursing or planning a pregnancy.
* Be a woman of childbearing potential who is not using an acceptable means of birth control
* Have a known allergy and/or sensitivity to the test article or its components.
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Have used an investigational drug or device within 30 days of Visit 1
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Inferior Corneal Fluorescein Staining Using The Ora Calibra Scale | Day 85
  An assessment of corneal fluorescein staining using the 0 [none] to 4 [worst] Ora Calibra Scale prior to and following exposure to a challenge in a controlled adverse environment (CAE)
Ocular Discomfort Using The Ora Calibra Scale | Day 85
  A patient-reported subjective assessment of ocular discomfort using the 0 [none] to 4 [worst] Ora Calibra Scale recorded at each study visit throughout the treatment period

SECONDARY OUTCOMES:
Corneal Fluorescein Staining Using The Ora Calibra Scale | 12 weeks
  An assessment of corneal fluorescein staining using the 0 [none] to 4 [worst] Ora Calibra Scale prior to and following exposure to a challenge in a controlled adverse environment (CAE)
Conjunctival Lissamine Green Staining Using The Ora Calibra Scale | 12 weeks
  An assessment of conjunctival lissamine green staining using the 0 [none] to 4 [worst] Ora Calibra Scale prior to and following exposure to a challenge in a controlled adverse environment (CAE)
Conjunctival Redness Using The Ora Calibra Scale | 12 weeks
  An assessment of conjunctival redness using the 0 [none] to 4 [worst] Ora Calibra Scale prior to and following exposure to a challenge in a controlled adverse environment (CAE)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Vita Eye Clinc, Shelby, North Carolina
  - Total Eye Care, P.A., Memphis, Tennessee

REFERENCES:
- [Derived] Evans D, Kenyon K, Ousler G, Watson M, Vollmer P, McLaurin EB, Torkildsen G, Winters J, Dodd J, Jordan R, Wills ST, Spana C. Efficacy and Safety of the Melanocortin Pan-Agonist PL9643 in a Phase 2 Study of Patients with Dry Eye Disease. J Ocul Pharmacol Ther. 2023 Nov;39(9):600-610. doi: 10.1089/jop.2023.0056. Epub 2023 Sep 7. PMID 37677000